CLINICAL TRIAL: NCT01929980
Title: Use of Bortezomib to Treat Refractory Autoimmune Cytopenia(s) in Allogeneic Stem Cell Transplantation
Brief Title: Bortezomib to Treat Significant Complication of HSCT
Acronym: Bortezomib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012:1089; NCT01930253 (obsolete NCT alias)
Record Dates: First submitted 2013-08-23; First posted 2013-08-28 (Estimated); Results first posted 2016-10-24 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Allogeneic Stem Cell Transplantation; Refractory Autoimmune Cytopenia(s)
Keywords: HSCT; cytopenia; immune suppression; proteasome inhibitor
MeSH Terms: conditions — Cytopenia | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bortezomib (Experimental): Four doses of bortezomib, 1.3mg/m2, will be given intravenously (through a needle in a vein) or subcutaneously (under the skin) on Days 1, 4, 8, 11.
  The format of receiving medications is- Therapy Dose and Route Frequency Rituximab 375 mg/m2 intravenously Once on day 1. Plasmapheresis 2 hours prior to Bortezomib Day 1,4, 8 and 11 Bortezomib 1.3 mg/m2 intravenously Day 1,4,8 and 11
  Interventions: Drug: Bortezomib

INTERVENTIONS:
Drug: Bortezomib
  Other Names: PS-341; Velcade

SUMMARY:
The purpose of this trial is to study the safety and effectiveness of a drug called Bortezomib for the treatment of low blood cell counts after bone marrow transplant.

DETAILED DESCRIPTION:
The purpose of this research study is to study the safety and effectiveness of a drug called bortezomib for the treatment of autoimmune cytopenia(s) (low blood cell counts) after bone marrow transplant that are not responding to standard treatments. Autoimmune cytopenias are low blood counts due to antibodies or proteins produced against an individual's own blood cells. Having a low red blood cell count (anemia) can make a person feel tired and require blood transfusions frequently. A low platelet count (blood cells that help blood to clot) can make a person bleed or bruise easily. A low neutrophil (white blood cell) count can make a person have infections.

All of these things can be a serious complication after bone marrow transplant and can cause prolonged hospital stay. Bortezomib is being used in children with certain types of blood cancer, however, bortezomib has not been used in children with autoimmune cytopenia(s) and its use in this study is investigational.

ELIGIBILITY:
Inclusion Criteria:

* All patients, having undergone allogeneic stem cell transplantation at our center.
* Should have failed at least 2 standard treatments for autoimmune cytopenias. Standard treatments include corticosteroids, rituximab, IVIG, plasmapheresis, withdrawal of cyclosporine, cyclophosphamide and MMF. Definition of "failed" treatment will be no response of cytopenia after 2 weeks of continued treatment OR requirement of daily GCSF at 10 mcgs/kg/day for autoimmune neutropenia despite 2 weeks of treatment, transfusions of packed red blood cells or platelets 3 times weekly for 2weeks despite continued treatment OR 5days/week plasmapheresis for 2 weeks and inability to wean the duration.
* Definition of autoimmune hemolytic anemia- development of anemia, where there is a hemoglobin drop of >2 g/dL/48 hours or an absolute value of hemoglobin < 8 g/dL, and evidence of hemolysis by positive direct Coombs test with compatible peripheral blood cell morphology, reticulocyte count and bilirubin level.
* Definition of autoimmune neutropenia - absolute neutrophil counts < 500 for 2 weeks and presence of anti-neutrophil antibodies.
* Definition of autoimmune thrombocytopenia- Platelet counts < 20,000 cells/uL for 2 weeks and presence of anti-platelet antibodies.

Exclusion Criteria:

* Ongoing life threatening infections
* Documented anaphylaxis to bortezomib
* Failed engraftment
* Relapse of primary malignancy
* ≥6/8 matched or haploidentical transplants

Ages: 4 Months to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2012-07; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Filipovich, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Bortezomib: Four doses of bortezomib, 1.3mg/m2, will be given intravenously (through a needle in a vein) or subcutaneously (under the skin) on Days 1, 4, 8, 11.
  The format of receiving medications is- Therapy Dose and Route Frequency Rituximab 375 mg/m2 intravenously Once on day 1. Plasmapheresis 2 hours prior to Bortezomib Day 1,4, 8 and 11 Bortezomib 1.3 mg/m2 intravenously Day 1,4,8 and 11
  Bortezomib
Period: Overall Study
Arm/Group | Bortezomib
Started | 4
Completed | 3
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bortezomib
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Response
Description: For Autoimmune Hemolytic Anemia- At least 3 of 5 criteria should be met.
  1. Stabilization of hemoglobin without transfusions by 2 weeks
  2. Conversion of DAT from + to - by 6 weeks
  3. Normalization of serum haptoglobin levels by 6 weeks
  4. Normalization of indirect bilirubin levels by 6 weeks
  5. Reduction in the frequency of transfusions by 50% by 4 weeks
  For Autoimmune Neutropenia- At least 2 of 3 criteria should be met.
  1. Stabilization of absolute neutrophil count by 2 weeks
  2. Undetectable antineutrophil antibodies by 6 weeks
  3. Reduction in GCSF dose by 50% by 6 weeks
  For Autoimmune Thrombocytopenia- At least 2 of 3 criteria should be met.
  1. Stabilization of platelet count without platelet transfusions by 2 weeks
  2. Undetectable antiplatelet antibodies by 6 weeks
  3. Reduction in the frequency of platelet transfusions by 50% from pre-bortezomib values by 6 weeks
Time Frame: 6 weeks
Measure: Number; unit: participants
Arm/Group | Bortezomib
Number analyzed (Participants) | 4
participants
  Neutropenia (n=3) | 3
  Thrombocytopenia (n=2) | 2
  Hemolytic Anemia (n=1) | 1

ADVERSE EVENTS:
Arm/Group | Bortezomib
Serious Adverse Events (participants affected / at risk) | 2/4
Other Adverse Events (participants affected / at risk) | 1/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bortezomib (N=4)
Pneumatosis Coli (Gastrointestinal disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
C diff colitis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bortezomib (N=4)
Nausea (Gastrointestinal disorders) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) — Cellulitis at subcutaneous injection site

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes